CLINICAL TRIAL: NCT01479322
Title: Correlation Between Hyperghrelinemia and Carotid Artery Intima-Media Thickness in Children With Prader-Willi Syndrome
Brief Title: Plasma Adiponectin Level and Vascular Endothelial and Smooth Muscle Cell Function in Children With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2006-11-056
Record Dates: First submitted 2011-07-31; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Prader-Willi Syndrome; Obesity
Keywords: Intima-media thickness; Ghrelin; Prader-Willi syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Context: Prader-Willi syndrome (PWS) is a genetic disorder characterized by childhood-onset obesity and endocrine dysfunction that leads to cardiovascular disability and early death within the first 3 decades of life.

Objectives: To assess the significance of risk factors for future disabilities, carotid artery intima-media thickness (IMT) was measured and correlated with known atherosclerotic risk factors in 27 children with PWS and 24 age-, sex-, and body mass index (BMI)-adjusted controls.

DETAILED DESCRIPTION:
Main outcome measures: Correlation of IMT with age, standard deviation score of BMI (BMI-SDS), high-density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL), C-reactive protein, HOMA-IR and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* obesity with PWS

Exclusion Criteria:

* chronic disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators studied twenty-seven children with PWS and 24 normal control subjects. The groups were adjusted for age, sex, and BMI.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, M.D, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine